CLINICAL TRIAL: NCT04385537
Title: The Ability of Pecan Consumption to Improve Vascular Function and Reduce Chronic Disease Risk in Aging Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Collaborators: American Pecan Council (Other)
Responsible Party: Principal Investigator, Jamie Cooper, PhD, Associate Professor, Dept. of Foods and Nutrition, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PROJECT00001978
Record Dates: First submitted 2020-04-30; First posted 2020-05-13 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Participants in this group avoid all nuts for 4-weeks
- PECAN (Experimental): Participants in this group consume 68 g of pecans/d with no other changes to their habitual diet and avoid all other nuts.
  Interventions: Dietary Supplement: PECAN

INTERVENTIONS:
Dietary Supplement: PECAN — Raw pecan halves without other changes to their habitual diet.
  Arms: PECAN

SUMMARY:
Background: To date, there are no published studies on the effects of pecans on vascular function following a high-fat meal.

Purpose: To examine the impact of daily pecan consumption for a 4-week period on vascular health and other markers of cardiovascular disease risk in aging adults.

DETAILED DESCRIPTION:
This will be a randomized, controlled trial in men and postmenopausal women (50-75y). Subjects will be randomized into one of the two study groups: a control group (CON) following their usual diet, or intervention group (PECAN) following their usual diet but also consuming 68g/day of pecans as a snack.

There will be 3 visits: A Screening visit and a baseline and post-diet intervention visit (4-weeks). Anthropometrics, questionnaires, a fasting blood sample, and fasting vascular measures will be collected at each visit. Subjects will participate in a saturated fatty acid meal challenge in which additional blood, vascular measurements will be collected.

Hypothesis: Daily pecan consumption will result in improved fasting blood lipids, vascular measures, antioxidant status, and appetite compared to the control group. Additionally, also the PECAN group will result in improved postprandial blood lipids and vascular measures compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Men and postmenopausal women (without menses for 1 yr and follicle stimulating hormone > 30 IU/mL) between the ages of 50-75y
* Body mass indexes (BMI) between 18-34.9kg/m2

Exclusion Criteria:

* Nut consumption >2 servings/week or tree nut butter consumption >3 servings/week
* Pre-menopausal and menopausal women, hormone replacement therapy if less than 2 years
* Regularly exercise more than 3 h/week
* Weight gain or loss more than 5% of their body weight in the past 3 months
* Plans to begin a weight loss/exercise regimen during the trial
* Gastrointestinal surgeries, conditions or disorders
* History of medical or surgical events that could affect swallowing
* Chronic or metabolic diseases
* Previous MI, stroke, or cancer
* Fasting blood glucose levels greater than 126 mg/dL
* Blood pressure greater than 180/120 mmHg
* Medication use affecting digestion and absorption, metabolism
* Lipid-lowering medications
* Medications for diabetes, depression, or ADD/ADHD
* Regular use of medications known to affect endothelial function or blood vessel tone
* Blood pressure medication and steroid/hormone therapies
* Individuals on a medically prescribed or special diet
* Individuals with food allergies to foods specifically in the study
* Excessively use alcohol (greater than 3 drinks/d for men; greater than 2 drinks/d for women)
* Tobacco or nicotine use
* Individuals taking fish oil and omega-3 fatty acid supplements
* Significant head trauma or brain surgery
* A score >26 on the Beck's Depression Inventory II (BDI-II)
* A score <24 on the Mini-Mental State Examination (MMSE) will be excluded.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2022-04-16 (Actual); Study Completion 2022-04-16 (Actual)

PRIMARY OUTCOMES:
Change in fasting and postprandial Flow-Mediated Dilation from baseline to 4 weeks | Baseline and 4 weeks
  Flow-Mediated Dilation %
Change in fasting and postprandial vessel diameter from baseline to 4 weeks | Baseline and 4 weeks
  baseline diameter (mm) and peak dilation (mm)
Change in fasting and postprandial reactive hyperemia velocity from baseline to 4 weeks | Baseline and 4 weeks
  Baseline velocity (cm/s) and reactive hyperemia velocity (cm/s)
Change in fasting and postprandial shear rate from baseline to 4 weeks | Baseline and 4 weeks
  baseline shear rate (sec.-1) and reactive hyperemia shear rate (sec.-1)
Change in fasting and postprandial Continuous-Wave Near-Infrared Spectrometry from baseline to 4 weeks | Baseline and 4 weeks
  O2 desaturation rate (%.sec-1), and O2 resaturation rate (%.sec-1)

SECONDARY OUTCOMES:
Change in fasting blood lipids from baseline to 4 weeks | Baseline and 4 weeks
  Total cholesterol (mg/dL), high-density lipoprotein (HDL) cholesterol (mg/dL), triglycerides (mg/dL), low-density lipoprotein (LDL) cholesterol (mg/dL), apolipoprotein B (mg/dL)
Change in baseline weight at 4 weeks | Baseline and 4 weeks
  weight (kg)
Change in baseline waist and hip circumference | Baseline and 4 weeks
  waist and hip circumference (cm)
Change in blood pressure from baseline to 4 weeks | Baseline and 4 weeks
  Systolic and Diastolic Blood Pressure (mm Hg)
Change in baseline total body fat percentage at 4 weeks | Baseline and 4 weeks
  total body fat percentage (%)
Change in fasting and postprandial insulin from baseline to 4 weeks | Baseline and 4 weeks
  Insulin (uU/mL)
Change in fasting and postprandial antioxidants from baseline to 4 weeks | Baseline and 4 weeks
  Total antioxidant capacity (uM trolox equivalents) measured via Oxygen Radical Absorbance Capacity (ORAC)
Change in fasting and postprandial lipid peroxidation from baseline to 4 weeks | Baseline and 4 weeks
  Malondialdehyde (MDA) (uM) measured via Thiobarbituric acid reactive substances (TBARS) assay.
Change in fasting inflammation from baseline to 4 weeks | Baseline and 4 weeks
  Interleukin-6 (pg/mL), C-reactive Protein (pg/mL), Tumor Necrosis Factor-α (pg/mL), Plasminogen Activator-1 (pg/mL)
Change in fasting and postprandial glucose and triglycerides from baseline to 4 weeks | Baseline and 4 weeks
  Glucose (mg/dL) and triglycerides (mg/dL)
Change in fasting and postprandial peptide YY, cholecystokinin (CCK), and ghrelin from baseline to 4 weeks | Baseline and 4 weeks
  Peptide YY (pg/mL), CCK (pg/mL), ghrelin (pg/mL)
Change in fasting and postprandial non-esterified free fatty acids (NEFA) from baseline to 4 weeks | Baseline and 4 weeks
  NEFA (mEq/L)
Change in fasting and postprandial hunger and satiety from baseline to 4 weeks | Baseline and 4 weeks
  Hunger, fullness, prospective consumption, and desire to eat measured via a Visual Analog Scale (VAS) (mm). The range of scores on the continuous VAS is between 0mm (no hunger, fullness, prospective consumption and desire to eat) and 100mm (the greatest feeling of hunger, fullness, prospective consumption and desire to eat)

OTHER OUTCOMES:
Change in fasting and postprandial composite cognitive function from baseline to 4 weeks | Baseline and 4 weeks. Measured at fasting, and 30 minutes and 3.5 hours postprandial.
  NIH tool box- Cognitive Battery (NIHTB-CB) computed- theta score for the sum of all subtests
Change in fasting and postprandial Cognitive Battery Motivation from baseline to 4 weeks | Baseline and 4 weeks. Measured at fasting, and 30 minutes and 3.5 hours postprandial.
  Visual Analogue Scale (VAS) (mm). This continuous scale is anchored by either no motivation (0mm) or extremely motivated (100mm).
Change in fasting and postprandial NIHTB-CB Flanker Inhibitory Control and Attention Test, and Dimensional Change Card Sort Test from baseline to 4 weeks | Baseline and 4 weeks. Measured at fasting, and 30 minutes and 3.5 hours postprandial.
  NIHTB-CB computed scores ranging from 0-10; high score representing greater accuracy
Change in fasting and postprandial NIHTB-CB Auditory Learning Test, Picture Sequence Memory Task and List Sorting Working Memory Test from baseline to 4 weeks | Baseline and 4 weeks. Measured at fasting, and 30 minutes and 3.5 hours postprandial.
  NIHTB-CB computed scores representing the number of correctly recalled items; higher scores indicating better memory.
Change in Pittsburg Sleep Quality Index scores from baseline to 4 weeks | Baseline and 4 weeks
  The scoring is out of 21 points, where a high score indicates poor sleep quality.
Change in State Trait Anxiety Inventory scores from baseline to 4 weeks | Baseline and 4 weeks
  The scoring is out of 80 points, where high score indicates higher levels of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Georgia- Department of Foods and Nutrition, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
The plan is to share group averages through publication.

REFERENCES:
- [Derived] Cogan B, Pearson RC, Jenkins NT, Paton CM, Cooper JA. A 4-Week Pecan-Enriched Diet Improves Postprandial Lipid Peroxidation in Aging Adults. J Med Food. 2023 Sep;26(9):654-662. doi: 10.1089/jmf.2023.0036. Epub 2023 Aug 28. PMID 37638838
- [Derived] Cogan B, Pearson RC, Jenkins NT, Paton CM, Cooper JA. A pecan-enriched diet reduced postprandial appetite intensity and enhanced peptide YY secretion: A randomized control trial. Clin Nutr ESPEN. 2023 Aug;56:25-35. doi: 10.1016/j.clnesp.2023.05.002. Epub 2023 May 8. PMID 37344080
- [Derived] Cogan B, Pearson RC, Paton CM, Jenkins NT, Cooper JA. Pecan-enriched diet improves cholesterol profiles and enhances postprandial microvascular reactivity in older adults. Nutr Res. 2023 Mar;111:44-58. doi: 10.1016/j.nutres.2023.01.001. Epub 2023 Jan 31. PMID 36822079